CLINICAL TRIAL: NCT00220766
Title: IGIV-C 10% Rapid Infusion Trial in Primary Immune Deficient Patients
Brief Title: Rapid Infusion of Immune Globulin Intravenous (Human) In Primary Immunodeficiency Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Gerald Klein, MD, Chief Medical Officer, Vice President of Medical and Clinical Affairs, Talecris Biotherapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 100348
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Immunologic Deficiency Syndrome; Agammaglobulinemia; Severe Combined Immunodeficiency; Wiskott-Aldrich Syndrome; Common Variable Immunodeficiency
Keywords: Primary Immune Deficiency; IGIV; Immunoglobulin G
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Agammaglobulinemia; Severe Combined Immunodeficiency; Wiskott-Aldrich Syndrome; Common Variable Immunodeficiency; Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Caprylates; Immunoglobulins, Intravenous; Glucose; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Infusion #1 (Week 0)Dextrose (0.14 mL/kg/min), then IGIV-C, 10% (0.08 mL/kg/min) ; Infusion #2 (Week 3-4)Dextrose (0.08 mL/kg/min), then IGIV-C, 10% (0.14 mL/kg/min)
  Interventions: Drug: Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified; Drug: Dextrose, 5% in Water
- Group 2 (Experimental): Infusion #1 (Week 0)Dextrose (0.08 mL/kg/min), then IGIV-C, 10% (0.14 mL/kg/min); Infusion #2 Dextrose (0.14 mL/kg/min), then IGIV-C, 10% (0.08 mL/kg/min)
  Interventions: Drug: Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified; Drug: Dextrose, 5% in Water

INTERVENTIONS:
Drug: Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified
  Other Names: Gamunex; IGIVnex; Gaminex; IGIV-C; Immune Globulin Intravenous (Human) , 10%; IGIV; BAY 41-1000; TAL-05-00004
Drug: Dextrose, 5% in Water

SUMMARY:
The objective of this study is to determine if the safety and tolerability of Immune Globulin Intravenous (Human), 10% caprylate/chromatography (IGIV-C)purified is similar when infused at two different infusion rates. The primary objective is to compare the incidence and severity of all infusion related adverse events when IGIV-C, 10% is administered at a rate of 0.14 mL/kg/min compared to a rate of 0.08 mL/kg/min after a single daily infusion.

DETAILED DESCRIPTION:
This is a prospective, single blind, randomized, multi-center cross-over trial in patients with Primary Immune Deficiency. Patients with a confirmed diagnosis of primary Immune Deficiency will be treated with two daily infusions given 3-4 weeks apart at the fixed individual IGIV dose regimen (400-600 mg/kg) established prior to entry into the study. Any subject with an established dose in the range of 200-399 mg/kg will be assigned to receive 400 mg/kg during the course of the study during the same dosing schedule established prior to entry into the study.

After a screening period lasting not more than four weeks, patients will be randomized into one of two cross-over groups. Patients randomized to Group 1 will receive their first IGIV-C, 10% dose at a rate of 0.08 mL/kg/min and their second infusion at a rate of 0.14 mL/kg/min, whereas patients randomized to Group 2 will receive IGIV-C, 10% at a rate of 0.14 mL/kg/min on the first infusion day and then 0.08 mL/kg/min on the second infusion day. All patients just prior to each IGIV-C, 10% infusion will receive the same volume of 5% dextrose as calculated for their IGIV-C, 10% infusion and given at a target rate according to the schema below.

Group 1:

* Infusion #1 (Week 0)Dextrose (0.14 mL/kg/min), then IGIV-C, 10% (0.08 mL/kg/min)
* Infusion #2 (Week 3-4)Dextrose (0.08 mL/kg/min), then IGIV-C, 10% (0.14 mL/kg/min)

Group 2:

* Infusion #1 (Week 0)Dextrose (0.08 mL/kg/min), then IGIV-C, 10% (0.14 mL/kg/min)
* Infusion #2 Dextrose (0.14 mL/kg/min), then IGIV-C, 10% (0.08 mL/kg/min)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary immune deficiency and medical records available for retrospective review for at least 3 months prior to entry into the trial
* Signed an informed consent written informed consent prior to initiation of any study related procedures
* Receiving regular infusions of IGIV at a fixed interval and dosage (in the range of 200-600 mg/kg given every 3-4 weeks) for at least three months prior to entry into the trial. Patients who are currently receiving less than 400 mg/kg are eligible for this trial and will be at the time of study enrollment be treated at 400 mg/kg

Exclusion Criteria:

* History or suspicion of significant allergic reaction to intravenous immune globulin, and/or blood products
* Documented history of selective IgA deficiency (serum level <5.0 mg/dL) and known antibodies to IgA
* Isolated IgG subclass deficiency with a normal total serum IgG level
* Other conditions which may interfere with the trial, include the patients demeanor or mental ability to follow instruction.
* Pretreatment with anti-pyretics or anti-histamines
* Congestive heart failure (New York Heart Association stage greater than Class II)
* Renal insufficiency (creatinine >2.5 mg/dL)
* Conditions whose symptoms and effects could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome)
* Pretreatment routinely required to control/ameliorate IGIV infusion-related adverse events (AEs)
* Any patient who requires IGIV dosing more frequently than every 3 weeks to maintain adequate trough levels
* Women of child bearing potential who do not practice adequate contraception (i.e. chemical or mechanical methods) and pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-08; Primary Completion 2002-08 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Infusion related adverse events | within 72 hours after infusion

SECONDARY OUTCOMES:
All adverse events | within 72 hours after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Gelfand, MD, Principal Investigator — National Jewish Medical and Research Center, Denver, CO
Locations (13):
- United States (9):
  - Departments of Medicine and Microbiology, Birmingham, Alabama
  - National Jewish Medical and Researach Center, Denver, Colorado
  - International Center for Interdisciplinary Studies of Immunology, Washington D.C., District of Columbia
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - University of South Florida College of Medicine, St. Petersburg, Florida
  - The Clinical Trials Center, Children's Hospital, New Orleans, Louisiana
  - Allergy, Asthma, and Immunology, Omaha, Nebraska
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Optimed Research, LLC, Columbus, Ohio
- Canada (4):
  - 3031 Hospital Drive Northwest, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Saint Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario